CLINICAL TRIAL: NCT02366468
Title: A 12-months, Randomized, VA-assessor Blinded, Multicenter, Controlled Phase IV Trial to Investigate Noninferiority of Two Treatment Algorithms (Discretion of the Investigator vs. Pro re Nata) of 0.5 mg Ranibizumab in Patients With Visual Impairment Due to Diabetic Macula Edema
Brief Title: Study of Efficacy of Ranibizumab in Different Regimens in Patients With Diabetic Macula Edema
Acronym: DIVERSE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRFB002DDE26; 2014-002854-37 (EudraCT Number)
Record Dates: First submitted 2015-01-12; First posted 2015-02-19 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetic macular edema; Visual impairment
MeSH Terms: conditions — Diabetic Retinopathy; Vision Disorders | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Discretion of the investigator (DI) (Experimental): ranibizumab 0.5 mg, after initial monthly treatment until maximum BCVA and no signs or no further change of disease activity, the investigator treated patients at their own discretion. There were no strict recommendations for retreatment or scheduling of upcoming visits.
  Interventions: Drug: ranibizumab 0.5 mg
- Pro re nata (PRN) (Active Comparator): ranibizumab 0.5 mg, after initial monthly therapy until maximum BCVA and no signs or no further improvement of disease activity, patients were monitored every month and retreated if any signs of disease activity occurred
  Interventions: Drug: ranibizumab 0.5 mg

INTERVENTIONS:
Drug: ranibizumab 0.5 mg — intravitreal injection
  Other Names: Lucentis

SUMMARY:
The purpose of this study was to demonstrate that the change of best corrected visual acuity (BCVA) was comparable in patients treated with ranibizumab at the discretion of the investigator vs. treatment according to a standard of care scheme (pro re nata, as needed).

ELIGIBILITY:
Inclusion Criteria:

* Patients with Type 1 or Type 2 diabetes mellitus with glycosylated hemoglobin (HbA1c) ≤ 12.0%
* Patients with visual impairment due to DME in at least one eye
* BCVA ≥ 24 and ≤ 78 letters in the study eye

Exclusion Criteria:

* Active intraocular inflammation
* Any active infection in either eye at the
* Structural damage within 0.5 disc diameter of the center of the macula in the study eye
* Uncontrolled glaucoma in either eye at screening

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2015-02-23 (Actual); Primary Completion 2017-06-08 (Actual); Study Completion 2017-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (25):
- Germany (25):
  - Novartis Investigative Site, Ahaus
  - Novartis Investigative Site, Bayreuth
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Bonn
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Freiburg I. Br
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Greifswald
  - Novartis Investigative Site, Halle
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hösbach
  - Novartis Investigative Site, Kempten
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Ludwigshafen
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Marburg
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Tübingen
  - Novartis Investigative Site, Ulm
  - Novartis Investigative Site, Würzburg

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: a total of 135 patients were randomized and assigned in a 1:1 ratio to the treatment arms.
Pre-assignment Details: At Screening, the eligibility criteria were performed.
Groups:
- Discretion of the Investigator (DI): Investigational - ranibizumab 0.5 mg
- Pro re Nata (PRN): Standard of Care - ranibizumab 0.5 mg
Period: Overall Study
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN)
Started (Randomized Safety Set) | 68 | 67
Full Analysis Set (FAS) (Randomized patients who received study treatment and had post-baseline primary endpoint assessments) | 67 | 66
Per Protocol Set (PPS) (All patients in the FAS who completed the trial without major protocol deviations) | 62 | 61
Completed | 62 | 58
Not Completed | 6 | 9
Not completed — Adverse Event | 2 | 0
Not completed — Withdrawal by Subject | 1 | 5
Not completed — Lost to Follow-up | 2 | 0
Not completed — Death | 1 | 2
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS). All patients randomized who received at least one application of study treatment and had at least one post-baseline assessment for the primary endpoint (BCVA).
Groups:
- Total: Total of all reporting groups
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN) | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: FAS
  years | 62.6 (13.73) | 65.0 (10.37) | 63.8 (12.19)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: FAS
  Participants
    Female | 22 | 25 | 47
    Male | 45 | 41 | 86
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 64 | 64 | 128
  Black | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Mean Average Change From Baseline in Best Corrected Visual Acuity (BCVA) of the Study Eye From Month 1 to Study Treatment Completion (Month 12)
Description: BCVA was assessed as letters read using Early Treatment Diabetic Retinopathy Study (ETDRS) charts. The mean average change from baseline was defined as the difference between the average level of BCVA (ETDRS letters) over all post-baseline assessments from Month 1 to Month 12. A positive change represents an improvement in visual acuity
Time Frame: Baseline, Month 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
Population: FAS - Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN)
Number analyzed (Participants) | 67 | 66
Letters
  Baseline (Day 1) | 67.4 (9.52) | 65.1 (9.59)
  post baseline average over month 1 to month 12 | 73.5 (9.50) | 73.8 (7.75)
  Visit-averaged change from baseline | 6.1 (6.54) | 8.6 (6.45)
Statistical Analysis 1: Comparison: Discretion of the Investigator (DI) vs Pro re Nata (PRN); The primary objective was to demonstrate that the mean visit-averaged change from baseline of BCVA over month 1 to treatment completion for the DI arm was non-inferior to the PRN arm; Test type: Non-Inferiority — non-inferiority margin: -4 letters; p = 0.002, ANCOVA; including study treatment (DI, PRN) and center as factors and baseline BCVA as continuous covariate; Median Difference (Final Values) = -0.9, 95% CI 2-sided [-3.04 to 1.27]

2. Secondary Outcome: Number of Visits
Description: Mean number of visits during the study
Time Frame: Baseline to Month 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Visits
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN)
Number analyzed (Participants) | 67 | 66
Visits | 12.7 (1.92) | 12.9 (2.25)

3. Secondary Outcome: Number of Injections
Description: mean number of injections in the study eye during the study
Time Frame: Baseline to Month 12
Population: FAS
Measure: Mean (Standard Deviation); unit: Injections
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN)
Number analyzed (Participants) | 67 | 66
Injections | 8.4 (2.98) | 7.8 (3.25)

4. Secondary Outcome: Number of Treatment Free Intervals
Description: A treatment-free interval is the interval between the first NO treatment given when the reason for NO treatment given is one of the three stability criteria and the first subsequent YES treatment given after that.
Time Frame: Baseline to Month 12
Population: FAS - including only patients with at least one treatment-free interval
Measure: Mean (Standard Deviation); unit: Intervals
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN)
Number analyzed (Participants) | 67 | 66
Intervals | 1.6 (0.76) | 1.7 (0.94)

5. Secondary Outcome: Mean Change in Central Subfield Retinal Thickness (CSRT)
Description: Evaluated by central reading center assessing OCT images
Time Frame: Baseline to Month 12
Population: FAS - Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN)
Number analyzed (Participants) | 67 | 66
μm
  Baseline | 420.0 (114.98) | 431.0 (128.13)
  Month 12 (LOCF) | 313.3 (61.21) | 320.6 (85.27)
  Change from Baseline to Month 12 (LOCF) | -106.7 (109.58) | -110.4 (101.97)
Statistical Analysis 1: Comparison: Discretion of the Investigator (DI) vs Pro re Nata (PRN); Test type: Superiority; p = 0.620, ANCOVA; containing the baseline values of the dependent variables as continuous covariates, and center and treatment as categorical covariates; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [-17.10 to 28.56]

6. Secondary Outcome: Mean Change of Foveal Center Point Thickness
Description: Evaluated by central reading center assessing OCT images
Time Frame: Baseline to Month 12
Population: FAS - LOCF - including only patients with assessments
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN)
Number analyzed (Participants) | 67 | 66
μm
  Baseline: number analyzed (Participants) | 64 | 60
  Baseline | 398.8 (144.10) | 405.0 (138.06)
  Month 12 - LOCF: number analyzed (Participants) | 64 | 60
  Month 12 - LOCF | 273.3 (84.85) | 280.6 (105.44)
  Change from Baseline to Month 12 (LOCF): number analyzed (Participants) | 64 | 60
  Change from Baseline to Month 12 (LOCF) | -125.6 (142.69) | -124.4 (113.29)
Statistical Analysis 1: Comparison: Discretion of the Investigator (DI) vs Pro re Nata (PRN); Test type: Superiority; p = 0.925, ANCOVA; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -1.5, 95% CI 2-sided [-33.66 to 30.59]

7. Secondary Outcome: Number of Participants With Change in Diabetic Retinopathy Study (DRS) Retinopathy Scale
Description: Evaluated by central reading center scoring fundus photography
Time Frame: Baseline to Month 12
Population: FAS - LOCF - including only patients with assessments
Measure: Count of Participants; unit: Participants
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN)
Number analyzed (Participants) | 67 | 66
Participants
  > 2 steps improvement | 7 | 7
  2 steps improvement | 3 | 4
  1 step improvement | 6 | 1
  0 steps | 38 | 34
  1 step loss | 4 | 4
  2 steps loss | 2 | 1
  > 2 steps loss | 1 | 5
  Missing | 6 | 10

ADVERSE EVENTS:
Time Frame: From start of study treatment until month 12
Arm/Group | Discretion of the Investigator (DI) | Pro re Nata (PRN)
All-Cause Mortality (participants affected / at risk) | 1/68 | 2/67
Serious Adverse Events (participants affected / at risk) | 13/68 | 22/67
Other Adverse Events (participants affected / at risk) | 44/68 | 43/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Discretion of the Investigator (DI) (N=68) | Pro re Nata (PRN) (N=67)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 1 | 1
Heart valve incompetence (Cardiac disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Eyelid function disorder (Eye disorders) | 0 | 1
Retinal detachment (Eye disorders) | 1 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 2
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Oedema peripheral (General disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Endophthalmitis (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1
VIIth nerve injury (Injury, poisoning and procedural complications) | 0 | 1
Blood glucose increased (Investigations) | 0 | 2
Urinary nitrogen increased (Investigations) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Balance disorder (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Diabetic neuropathy (Nervous system disorders) | 1 | 0
Facial paralysis (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diabetic foot (Skin and subcutaneous tissue disorders) | 1 | 1
Behcet's syndrome (Vascular disorders) | 1 | 0
Circulatory collapse (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 1
Hypertensive crisis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Discretion of the Investigator (DI) (N=68) | Pro re Nata (PRN) (N=67)
Cataract (Eye disorders) | 2 | 5
Conjunctival haemorrhage (Eye disorders) | 13 | 14
Corneal erosion (Eye disorders) | 4 | 4
Eye irritation (Eye disorders) | 1 | 5
Eye pain (Eye disorders) | 7 | 4
Foreign body sensation in eyes (Eye disorders) | 6 | 1
Macular oedema (Eye disorders) | 5 | 5
Ocular discomfort (Eye disorders) | 4 | 4
Visual acuity reduced (Eye disorders) | 7 | 8
Visual impairment (Eye disorders) | 4 | 2
Vitreous floaters (Eye disorders) | 3 | 5
Vitreous haemorrhage (Eye disorders) | 6 | 2
Conjunctivitis (Infections and infestations) | 1 | 4
Viral upper respiratory tract infection (Infections and infestations) | 19 | 18
Glycosylated haemoglobin increased (Investigations) | 5 | 7
Intraocular pressure increased (Investigations) | 8 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 1
Headache (Nervous system disorders) | 4 | 1
Haematoma (Vascular disorders) | 4 | 0
Hypertension (Vascular disorders) | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-04-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT02366468/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-13): https://cdn.clinicaltrials.gov/large-docs/68/NCT02366468/SAP_001.pdf